CLINICAL TRIAL: NCT05759767
Title: The Efficacy and Safety of Medical Expulsive Therapy After Extracorporeal Shock Wave Lithotripsy (ESWL) in Pediatric Urolithiasis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Ped MET SWL
Record Dates: First submitted 2023-02-26; First posted 2023-03-08 (Actual); Last update posted 2023-03-10 (Actual); Status verified 2023-02

CONDITIONS: Tamsulosin; Extracorporeal Shock Wave Lithotripsy; Stone, Kidney; Stone, Urinary; Pediatric Disorder
Keywords: Extracorporeal Shock Wave Lithotripsy; tamsulosin
MeSH Terms: conditions — Kidney Calculi; Urinary Calculi | interventions — Tamsulosin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tamsulosin (Active Comparator): Children in this group will receive medical expulsive therapy in the form of (tamsulosin at a dose of 0.01 mg/kg once daily for 3 weeks after ESWL session.
  Interventions: Drug: Tamsulosin
- Placebo (Placebo Comparator): Children in this group will receive Placebo for 3 weeks after ESWL session.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tamsulosin — Children in this group will receive medical expulsive therapy in the form of (tamsulosin at a dose of 0.01 mg/kg once daily for 3 weeks after ESWL session.
  Arms: Tamsulosin
Drug: Placebo — Children in this group will receive placebo once daily for 3 weeks after ESWL session.
  Arms: Placebo

SUMMARY:
The aim of this study is to evaluate the clinical efficacy and safety of MET after ESWL in pediatric urolithiasis.

ELIGIBILITY:
Inclusion Criteria:

* Radio- opaque renal stone ≤ 2 cm or ≤ 1cm lower calyceal stone
* Normal kidney function.

Exclusion Criteria:

* Bleeding diatheses
* Uncontrolled UTIs
* Severe skeletal malformations

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 120 (Estimated)
Dates: Start 2021-02-01 (Actual); Primary Completion 2023-12-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
assess the Stone-free rate (SFR) between groups | three months
  SFR is defined as complete stone removal without visible stone fragments on radiological studies assessed by Low dose Non Contrast Computed Tomography

CONTACTS AND LOCATIONS:
Locations (1):
- Urology and Nephrology Center, Al Mansurah, Egypt